CLINICAL TRIAL: NCT06095765
Title: Colchicine in Belgium in Patients With Coronary Artery Disease
Brief Title: Colchicine in Belgium in Patients With Coronary Artery Disease After Percutaneous Coronary Intervention
Acronym: COL BE PCI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: University Hospital, Ghent (Other); Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Principal Investigator, Ian Buysschaert, MD PhD, MD, PhD, Chief investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ONZ-2023-0237; KCE-INV-21-1324 (Other Grant/Funding Number: Belgian Health Care Knowledge Centre (KCE)); 2023-505028-74-00 (Other: EU CT number)
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; colchicine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine; Tablets

STUDY DESIGN:
Intervention Model Description: Colchicine versus placebo (1:1)
Who Masked: Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): Colchicine 0.5 mg oral once daily, in addition to SOC
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Placebo (Placebo Comparator): Placebo oral once daily, in addition to SOC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet — Oral intake of 0.5 mg colchicine once daily
  Arms: Colchicine
Drug: Placebo — Oral intake of matching placebo once daily
  Arms: Placebo

SUMMARY:
The main aim of this trial is to determine whether there are fewer cardiovascular events when patients with coronary artery disease take a low dose of colchicine of 0.5 mg daily on top of optimal standard treatment after treatment with PCI, compared with placebo in combination with optimal standard treatment. More specifically, we aim to investigate the benefits of a daily low dose of colchicine in patients with coronary artery disease after treatment with PCI, to confirm that a daily low dose of colchicine helps prevent additional incidents in coronary artery disease, and to identify a subgroup of patients with CAD who are at increased risk for cardiovascular events and could benefit most from colchicine.

DETAILED DESCRIPTION:
This is a prospective, randomised, double-blind, multicenter, placebo-controlled phase III pragmatic superiority trial comparing colchicine 0.5 mg with placebo administered orally once-daily in up to 2770 participants with CAD treated with PCI. Participants will be randomised in a 1:1 ratio to receive either colchicine 0.5 mg or placebo as an adjunct to standard of care. The trial is event driven with trial closure being performed when the targeted number of 566 primary endpoint events has been reached.

Participants will be seen by the site staff 1 month after randomisation and thereafter every 12 months as per standard of care (SOC) and for IMP dispense and compliance, completing questionnaires and outcome event assessment until end of study. After the first month, a telephone visit will be scheduled every 6 months in between two standard of care on-site visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥45 years.
2. Coronary artery disease treated with PCI and optimal medical therapy, with at least one additional risk factor (based on SMART):

   1. Age ≥ year
   2. Diabetes mellitus, on treatment or new diagnosis with HbA1c ≥6.5%
   3. Current smoking
   4. Treated hypertension or lood pressure systolic ≥ 4 mmHg or diastolic ≥ mmHg
   5. Total cholesterol >240 mg/dl untreated, or treated LDL >70 mg/dl
   6. HDL <40 mg/dl
   7. hsCRP >2 mg/L AND chronic coronary syndrome (CCS)
   8. eGFR <60 ml/min (MDRD)
   9. history of vascular disease:

      * CAD (PCI prior to index, CABG, MI)
      * stroke (ischemic or hemorrhagic)
      * carotid artery revascularisation
      * PAD (revascularisation, ABI <0.85 at rest, amputation due to atherosclerotic disease)
      * AAA (repair, distal aortic anteroposterior diameter >3.0cm)
3. Able to be enrolled/randomized between 2 hour and 5 days post PCI.
4. Written informed consent.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or of childbearing potential who are not using an effective method of contraception. Or women who intend to donate oocytes.
2. Men who plan to father children during the study period or who are unwilling to use effective forms of contraception. Or men who intend to donate sperm.
3. Any contraindication or known intolerance to colchicine.
4. Chronic use of -or need for- colchicine.
5. Auto-immune disease or other condition requiring current or planned chronic systemic steroids, immunosuppressant or biologic drug targeting the immune system (for example, TNF blockers, anakinra, rituximab, abatacept, tocilizumab etc.).
6. Creatinine clearance <30 mL/min/1.73 m2.
7. Cirrhosis Child-Pugh stadium B and C, or acute severe liver disease
8. Neuromuscular disease or non-transient CK levels > 5 x ULN (unless due to MI).
9. History of cancer or lymphoproliferative disease within the last 3 years, other than successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma, or localized cervix carcinoma in situ.
10. Current or planned use of any strong inhibitor of CYP3A4 or p-glycoprotein: macrolide antibiotics (clarithromycin, telithromycin), azole antifungal agents (ketoconazole, voriconazole, fluconazole, itraconazole), cyclosporine, HIV medication (ritonavir, lopinavir, tipranavir, atazanavir, darunavir, indinavir, saquinavir).
11. Chronic diarrhea, or inflammatory owel disease (Crohn's disease or ulcerative colitis).
12. Drug or alcohol abuse.
13. Planned cardiovascular intervention known on the day of screening.
14. Currently enrolled in another investigational trial.
15. Considered to be an unsuitable candidate by the investigator.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2770 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Time from randomisation to first occurrence of a composite endpoint consisting of: all-cause death, spontaneous (non-procedural) non-fatal myocardial infarction (Type 1, 4B & C), non-fatal stroke, or coronary revascularisation. | 44 months

SECONDARY OUTCOMES:
Time from randomisation to first occurrence of a composite of specific cardiovascular endpoints | 44 months
  Time from randomisation to first occurrence of a composite of: cardiovascular death, spontaneous (non-procedural) non-fatal myocardial infarction (Type 1, 4B & C), non-fatal stroke or coronary revascularisation
Time from randomisation to first occurrence of a composite of hard endpoints consisting of: all-cause death, spontaneous (non-procedural) non-fatal myocardial infarction (Type 1, 4B & C), non-fatal stroke | 44 months
Time from randomisation to first occurrence of breakdown components of primary endpoint and atherosclerosis-related diseases | 44 months
  Time from randomisation to first occurrence of: all-cause death, cardiovascular death, spontaneous (non-procedural) non-fatal myocardial infarction (Type 1, 4B & C), non-fatal stroke, coronary revascularisation, ischemia driven coronary revascularisation, stent thrombosis, peripheral artery revascularisation, transient ischemic attack (TIA) treated with carotid revascularisation
Time from randomisation to occurrence of first as well as recurrent endpoints consisting of: all-cause death, spontaneous (non-procedural) non-fatal myocardial infarction (Type 1, 4B & C), non-fatal stroke, or coronary revascularisation. | 44 months
Change from randomisation to year 1 and to end of study of participants reported outcomes (based on ICHOM Standard Set for CAD): Angina Frequency scale | 44 months
  Change from randomisation to year 1 and to end of study of participants reported outcomes:
  Seattle Angina Questionnaire (SAQ) Angina Frequency Scale: categorizes angina (chest pain) frequency as following: daily angina (score = 0-30), weekly angina (score = 31-60), monthly angina (score = 61-99), and no angina (score = 100). Higher score indicates better outcome.
Change from randomisation to year 1 and to end of study of participants reported outcomes (based on ICHOM Standard Set for CAD): Dyspnea | 44 months
  Change from randomisation to year 1 and to end of study of participants reported outcomes:
  Dyspnea (Rose Dyspnea Scale): a four-item questionnaire that assesses a patients' dyspnea level with common activities. One point is assigned to each activity associated with dyspnea. Scores range from 0 to 4. Higher score indicates worse outcome.
Change from randomisation to year 1 and to end of study of participants reported outcomes (based on ICHOM Standard Set for CAD): Depression. | 44 months
  Change from randomisation to year 1 and to end of study of participants reported outcomes:
  Depression (Patient Health Questionnaire PHQ-2): inquires about the frequency of depressed mood and anhedonia. Scores range from 0 to 6. Higher score indicates worse outcome.
Change from randomisation to year 1 and to end of study of participants reported outcomes (based on ICHOM Standard Set for CAD): Health-related quality of life. | 44 months
  EuroQol five dimensions five level (EQ-5D-5L): consists of a descriptive system of self-perceived health status along fve dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and a visual analogue scale (VAS) which provides a self-rating of the general health status on a scale from 0 (worst imaginable state of health) to 100 (best imaginable state of health).

OTHER OUTCOMES:
Change from randomisation to year 1 (and year 2 if available): in hsCRP as a measure of Inflammation. | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from:
  (high sensitivity) C-reactive protein (mg/dl)
Change from randomisation to year 1 (and year 2 if available): in white blood cell count as a measure of Inflammation. | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from:
  white blood cell count (/μl)
Change from randomisation to year 1 (and year 2 if available) in total cholesterol. | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from:
  total cholesterol (mg/dl)
Change from randomisation to year 1 (and year 2 if available) in low density lipoprotein. | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from:
  low density lipoprotein (LDL) (mg/dl)
Change from randomisation to year 1 (and year 2 if available) in high density lipoprotein . | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from:
  high density lipoprotein (HDL) (mg/dl)
Change from randomisation to year 1 (and year 2 if available) in triglycerides. | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from:
  triglycerides (mg/dl)
Change from randomisation to year 1 (and year 2 if available) in kidney function. | 24 months
  Change from randomisation to year 1 (and year 2 if available) in blood lab results from: estimated glomerular filtration rate (ml/min)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Buysschaert, MD, PhD, Principal Investigator — ian.buysschaert@azsintjan.be
Locations (19):
- Belgium (19):
  - Algemeen Stedelijk Ziekenhuis Campus Aalst, Aalst
  - Het Ziekenhuisnetwerk Antwerpen, Antwerp
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Imelda, Bonheiden
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Humani Charleroi, Charleroi
  - Grand Hôpital de Charleroi, Charleroi
  - Ziekenhuis Oost Limburg, Genk
  - AZ Sint-Lucas & Volkskliniek, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Algemeen Ziekenhuis Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - Centre Hospitalier Regional De La Citadelle, Liège
  - Clinique Saint-Luc Bouge, Namur
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
  - UCL Mont-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiolet ATL, Opstal TSJ, Mosterd A, Eikelboom JW, Jolly SS, Keech AC, Kelly P, Tong DC, Layland J, Nidorf SM, Thompson PL, Budgeon C, Tijssen JGP, Cornel JH. Efficacy and safety of low-dose colchicine in patients with coronary disease: a systematic review and meta-analysis of randomized trials. Eur Heart J. 2021 Jul 21;42(28):2765-2775. doi: 10.1093/eurheartj/ehab115. PMID 33769515
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Tong DC, Quinn S, Nasis A, Hiew C, Roberts-Thomson P, Adams H, Sriamareswaran R, Htun NM, Wilson W, Stub D, van Gaal W, Howes L, Collins N, Yong A, Bhindi R, Whitbourn R, Lee A, Hengel C, Asrress K, Freeman M, Amerena J, Wilson A, Layland J. Colchicine in Patients With Acute Coronary Syndrome: The Australian COPS Randomized Clinical Trial. Circulation. 2020 Nov 17;142(20):1890-1900. doi: 10.1161/CIRCULATIONAHA.120.050771. Epub 2020 Aug 29. PMID 32862667
- [Background] Dorresteijn JA, Visseren FL, Wassink AM, Gondrie MJ, Steyerberg EW, Ridker PM, Cook NR, van der Graaf Y; SMART Study Group. Development and validation of a prediction rule for recurrent vascular events based on a cohort study of patients with arterial disease: the SMART risk score. Heart. 2013 Jun;99(12):866-72. doi: 10.1136/heartjnl-2013-303640. Epub 2013 Apr 10. PMID 23574971
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Derived] De Cock E, Kautbally S, Timmermans F, Bogaerts K, Hanet C, Desmet W, Gurne O, Vranckx P, Hiltrop N, Dujardin K, Vanduynhoven P, Vermeersch P, Pirlet C, Hermans K, Van Reet B, Ferdinande B, Aminian A, Dewilde W, Guedes A, Simon F, De Roeck F, De Vroey F, Jukema JW, Sinnaeve P, Buysschaert I. Low-dose colchicine for the prevention of cardiovascular events after percutaneous coronary intervention: Rationale and design of the COL BE PCI trial. Am Heart J. 2024 Dec;278:61-71. doi: 10.1016/j.ahj.2024.08.022. Epub 2024 Sep 2. PMID 39233210